CLINICAL TRIAL: NCT02272686
Title: Targeting Bruton's Tyrosine Kinase (BTK) With Ibrutinib After Autologous Stem Cell Transplantation in "Double-Hit" B-Cell Lymphoma
Brief Title: Ibrutinib Post Stem Cell Transplantation (SCT) in Double-Hit B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0096; NCI-2015-00843 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Lymphoma
Keywords: Lymphoma; Blood And Marrow Transplantation; Post Autologous Stem Cell Transplantation; SCT; B-cell lymphoma; Ibrutinib; PCI-32765; Imbruvica
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib (Experimental): Ibrutinib started at a daily dose of 560 mg by mouth daily for up to 3 years.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — 560 mg by mouth daily.
  Other Names: PCI-32765; Imbruvica

SUMMARY:
The goal of this clinical research study is to learn if ibrutinib can help to control lymphoma in patients who have had an autologous stem cell transplant (a transplant using your own stem cells). The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

If you take part in this study, you will take ibrutinib by mouth 1 time each day for up to 3 years. You must swallow the capsules whole with a glass (about 8 ounces) of water. Do not open, break, or chew the capsules. You should take ibrutinib at the same time every day.

If you miss a dose of ibrutinib, take it as soon as you remember on the same day. Take your next dose of ibrutinib at your regular time on the next day. Do not take 2 doses of ibrutinib on the same day to make up for a missed dose.

You will be given a study drug diary to write down what time you take each dose of ibrutinib. You need to bring the study drug diary, any leftover study drug, and any empty study drug containers with you to each visit.

The dose of ibrutinib you receive may be lowered, if the doctor thinks it is needed.

Study Visits:

One (1) time during Weeks 1-4, 6, and 8 and then 1 time each month after that for up to 3 years after your first dose of ibrutinib, blood (about 2 tablespoons) will be drawn for routine tests and to check your kidney and liver function. The blood draws may be performed at MD Anderson or at a lab closer to your home.

If the study doctor thinks it is needed, you may need to have these blood draws more often.

Around 1 month after your first dose of ibrutinib, you will have a bone marrow biopsy/aspirate to check the status of the disease, if the study doctor thinks it is needed. To collect a bone marrow biopsy/aspirate, an area of the hip or other site is numbed with anesthetic, and a small amount of bone and bone marrow is withdrawn through a large needle.

Around 3, 6, 9, and 12 months, then every 6 months for 3 years after your first dose of ibrutinib:

* You will have a physical exam.
* You will have computed tomography (CT) scans to check the status of the disease.
* You will have a bone marrow biopsy/aspirate to check the status of the disease.

Length of Study:

You may continue taking the study drug for up to 3 years. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on this study will be over after about 3 years.

Follow-Up Visit:

You will continue to have the CT scans and blood draws described in the study visits section 1 time a year for up to 3 years.

If you had a positron emission tomography (PET) scan that was performed at the time of your transplant and the scan showed that the disease was still in your body, you will have a PET scan 1 time each year while taking ibrutinib. The PET scan will not be repeated if the results show that there is no disease in the body.

This is an investigational study. Ibrutinib is FDA-approved and commercially available for the treatment of many types of cancers, including mantle cell lymphoma with 1 prior therapy. The use of ibrutinib to treat double hit lymphoma after an autologous stem cell transplant is considered investigational. The study doctor can explain how the study drug is designed to work.

Up to 30 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed double hit in first complete remission, anytime during the first 3 months after chemoimmunotherapy followed by autologous stem cell transplantation if there was no evidence of progression.
2. Double hit lymphoma is defined as B-cell lymphoma with genetic abnormalities involving A) and in addition, B) and/or C): A) C-MYC arrangement or amplification by FISH study. B) BCL2 rearrangement or amplification by FISH study. C) BCL6 rearrangement or amplification by FISH study.
3. ANC >/= 1,000, platelets >/= 75,000.
4. AST and/or ALT < 3 times the ULN.
5. Creatinine clearance > 30 ml/min (Cockcroft-Gault formula using ideal body weight).
6. Male or female age >/= 18 years.
7. ECOG performance status </= 2.
8. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
9. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information.
10. Patient should preferably have received a pre-transplant conditioning with rituximab and Carmustine/Etoposide/Cytarabine/Melphalan/Rituxan (BEAM/R) . Other regimens which are similar may be accepted at the discretion of the PI.

Exclusion Criteria:

1. Prior chemotherapy within 3 weeks, nitrosoureas (carmustine) within 6 weeks, therapeutic anticancer antibodies within 4 weeks, radio- or toxin-immunoconjugates within 10 weeks, radiation therapy within 3 weeks, or major surgery within 2 weeks of first dose of study drug.
2. Relapsed within three months post transplant.
3. History of other malignancies within the past year except for treated basal cell or squamous cell skin cancer or in situ cervical cancer.
4. Known CNS lymphoma.
5. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
6. Requires treatment with a strong cytochrome P450 (CYP)3A inhibitor (i.e. Voriconazole, posaconazole, itraconazole, clarithromycin, etc.) or inducer (carbamazepine, rifampin, phenytoin, etc.).
7. AST and/or ALT >/= 3 times the ULN.
8. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or symptomatic ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
9. Known history of human immunodeficiency virus or active infection with hepatitis C virus or hepatitis B virus or any uncontrolled active systemic infection.
10. Positive pregnancy test in women of childbearing potential.
11. Lactating or pregnant or will not agree to use contraception during the study and for 30 days after the last dose of study drug if sexually active and able to bear children.
12. Concomitant use of warfarin or other Vitamin K antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issa F. Khouri, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 6/3/2016 to 2/21/2017.
Pre-assignment Details: Ibrutinib maintenance will not be started if patient relapses post transplant
Groups:
- Ibrutinib Maintenance: Ibrutinib maintenance after autologous stem cell transplantation (SCT) in double-hit lymphoma
Period: Overall Study
Arm/Group | Ibrutinib Maintenance
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib Maintenance
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: Participants will be assessed for disease status and survival.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib Maintenance
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Overall Survival (OS)
Description: Participants will be assessed at 3 year time point for survival.
Time Frame: Three Years
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib Maintenance
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: through study completion, an average of 10 months
Arm/Group | Ibrutinib Maintenance
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT02272686/Prot_SAP_000.pdf